CLINICAL TRIAL: NCT01054053
Title: Phase 3, Vaccinal Activity Assessment of MenBVac Against Nesseiria Menigitidis B:14,P1.7,16 Strain in Child.
Brief Title: Evaluation of Immune Response Against the Strain of Neisseria Meningitidis B: 14, P1-7, 16 Patients Have to be Vaccinated MenBVac®
Acronym: EFFIVAC
Status: Completed | Type: Observational
Sponsor: University Hospital, Rouen (Other)
Collaborators: Institut Pasteur (Industry)
Responsible Party: Sponsor
Other Study IDs: 2009/042/HP; 2009-011401-16
Record Dates: First submitted 2009-11-26; First posted 2010-01-22 (Estimated); Last update posted 2012-03-23 (Estimated); Status verified 2012-03

CONDITIONS: Vaccination
Keywords: Neisseria meningitidis B:14, P1-7, 16; Serum bactericidal activity; Menbvac

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood samples
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- 1: children born between 06/04/2004 and 17/04/2008 and called to menBvac vaccination and living around Neufchatel en Bray.

SUMMARY:
The main objective of the study is to estimate the proportion of children, born between the 06/04/2004 and the 17/004/2008, living around Neufchatel en Bray, vaccinated by MenBVac, with a serum bactericidal activity against B:14,P1-7,16 clone related to a protection (>= 4), before the first vaccination (T0), after the second MenBvac vaccination (6 weeks after the second vaccination), before the third MenBvac vaccination and after the third MenBvac vaccination (6 weeks after the second vaccination) and one year after the third menBvac vaccination.

ELIGIBILITY:
Inclusion Criteria:

* children born between 06/04/2004 and 17/04/2008, living in Neufchatel en Bray, vaccinated five times by MenBVac
* parental authority(ies)assent

Exclusion Criteria:

* no parental authority(ies)assent
* no blood sample during the third vaccination
* impossibility of third vaccination
* children with guardianship
* children yet vaccinated or non eligible for vaccination

Ages: 1 Year to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: children born between 06/04/2004 and 17/04/2008, living Neufchatel en bray.
Sampling Method: Non-Probability Sample
Enrollment: 218 (Actual)
Dates: Start 2009-04; Primary Completion 2010-10 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
assessment of natural Immunity with measure of percent of children who have hSBA title >= 4 at TO. assessment of antibodies blood persistence during measurement of percent of children who have hSBA title >= 4 | 18 months

CONTACTS AND LOCATIONS:
Locations (1):
- Maison Du Département, Neufchâtel-en-Bray, France